CLINICAL TRIAL: NCT00560443
Title: Randomized Controlled Trial on Effectiveness of Ketorolac and Tramadol in Not Compound Fractures of Child
Brief Title: RCT on Ketorolac and Tramadol in Bone Fractures Pain of Child
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RC 30/07
Record Dates: First submitted 2007-11-07; First posted 2007-11-19 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Fracture; Pain
Keywords: bone fracture; ketorolac; tramadol
MeSH Terms: conditions — Fractures, Bone; Pain | interventions — Ketorolac; Tramadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): children 4-17 y. old with not compound bone fracture treated with ketorolac
  Interventions: Drug: ketorolac
- 2 (Experimental): children 4-17 y. old with not compound bone fracture treated with tramadol
  Interventions: Drug: tramadol

INTERVENTIONS:
Drug: ketorolac — 0,5 mg/kg per os one time
  Arms: 1
Drug: tramadol — 2,5 mg/ kg per os in one dose
  Arms: 2

SUMMARY:
Randomized double blind Trial with the aim to estimate effectiveness of two therapeutic regimes per os on pain due to not compound bone fractures in child 4-17 years old:

* ketorolac 0,5 mg/kg (1 drop every 2 Kg)
* tramadol 2,5 mg/Kh (1 drop every 2 Kg)

Intensity of pain will be estimated with linear 1 to 10 or analogic McGrath type scale every 20 min.

The main objectives are the evaluation of pain decreasing in every group, the time of decreasing, the intensity of pain during procedures (ex. Xray) and the occurrence of side effects Secondary outcomes are comparison between the two groups on effectiveness on pain and on side effects

ELIGIBILITY:
Inclusion Criteria:

* Children 4-17 years old with not compound bone fracture presenting in emergency room

Exclusion Criteria:

* Compound fracture
* Occurring pain still treated
* Contraindicated ketorolac or tramadol use
* Informed consensus not obtained

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 133 (Actual)
Dates: Start 2008-02 (Actual); Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
estimation of pain reduction in every arm of the trial with linear 1-10 pain scale or for children 4 - 6 years old with analogic MacGrath type scale | 6 hours (or until the end of procedures)

SECONDARY OUTCOMES:
comparison between the two groups on effectiveness on pain, measured with linear and analogic scale (see above) | 6 hours or until the end of procedures

CONTACTS AND LOCATIONS:
Overall Officials: Edoardo Guglia, md, Principal Investigator — IRCCS Burlo Garofolo
Locations (1):
- IRCCS Burlo Garofolo, Trieste, Italy

REFERENCES:
- [Derived] Neri E, Maestro A, Minen F, Montico M, Ronfani L, Zanon D, Favret A, Messi G, Barbi E. Sublingual ketorolac versus sublingual tramadol for moderate to severe post-traumatic bone pain in children: a double-blind, randomised, controlled trial. Arch Dis Child. 2013 Sep;98(9):721-4. doi: 10.1136/archdischild-2012-303527. Epub 2013 May 23. PMID 23702435